CLINICAL TRIAL: NCT01694264
Title: A Randomized, Double-blinded, Phase 3, Multicenter, Investigator-initiated Trial for Entecavir for Prophylaxis of Hepatitis B Virus (HBV) Reactivation in HBV Surface Antigen or Anti-HBc Positive Patients Undergoing Anti-TNFα Treatment
Brief Title: Study of Anti-Viral Prophylaxis for HBsAg(+) or HBcAb(+)/HBsAb(-) Patients Starting Anti-TNFα
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Delayed recruitment, unable to meet calculated sample size
Sponsor: Seoul National University Hospital (Other)
Collaborators: Konkuk University Medical Center (Other); Kyungpook National University Hospital (Other); Kyunghee University Medical Center (Other); Kyung Hee University Hospital at Gangdong (Other); Gachon University Gil Medical Center (Other); Daegu Catholic University Medical Center (Other); Eulji University Hospital (Other); SMG-SNU Boramae Medical Center (Other); The Catholic University of Korea (Other); Severance Hospital (Other); Ajou University School of Medicine (Other); Ewha Womans University Mokdong Hospital (Other); Inha University Hospital (Other); Chonnam National University Hospital (Other); Chonbuk National University Hospital (Other); Chungnam National University Hospital (Other); Hallym University Medical Center (Other); Hanyang University (Other); Dong-A University (Other); Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Yeong-Wook Song, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H-1112-073-390
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Chronic Hepatitis B; Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis; Juvenile Idiopathic Arthritis
Keywords: HBV surface antigen; Anti-HBc positive; Anti-TNFα Treatment; Reactivation
MeSH Terms: conditions — Hepatitis B, Chronic; Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Arthritis, Juvenile | interventions — entecavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): Entecavir (Baraclude (Bristol-Myers Squibb) 0.5mg.) will be taken orally on an empty stomach (2 hours after a meal or at least 2 hours before the next meal), once daily from 1 week before starting anti-TNFα and continue 72 weeks after anti-TNFα is administered.
  Interventions: Drug: Entecavir
- Control Group (Placebo Comparator): Placebo of Entecavir (prepared by Bristol-Myers Squibb) will be taken orally on an empty stomach (2 hours after a meal or at least 2 hours before the next meal), once daily from 1 week before starting anti-TNFα and continue 72 weeks after anti-TNFα is administered.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Entecavir — Entecavir (Baraclude (Bristol-Myers Squibb) 0.5mg.) will be taken orally on an empty stomach (2 hours after a meal or at least 2 hours before the next meal), once daily from 1 week before starting anti-TNFα and continue 72 weeks after anti-TNFα is administered.
  Other Names: Baraclude (Bristol-Myers Squibb) 0.5mg
  Arms: Experimental Group
Drug: Placebo — Placebo of Entecavir (prepared by Bristol-Myers Squibb) will be taken orally on an empty stomach (2 hours after a meal or at least 2 hours before the next meal), once daily from 1 week before starting anti-TNFα and continue 72 weeks after anti-TNFα is administered.
  Other Names: placebo, prepared by Bristol-Myers Squibb
  Arms: Control Group

SUMMARY:
Analysis of effect of anti-TNFα treatment on HBV reactivation among patients with systemic rheumatic disease, especially rheumatoid arthritis

DETAILED DESCRIPTION:
Biologic agents, especially anti-TNFα treatments are widely used in inflammatory arthritis such as rheumatoid arthritis (RA) and ankylosing spondylitis (AS). More than 60% of RA or AS patients achieve good clinical response to anti-TNFα treatment. However, TNFα is also an important mediator participating in the normal immune response to infectious agents, in particular intracellular microorganisms in the human body. Therefore, opportunistic infections such as tuberculosis, viral and fungal infections have been of concern when using anti-TNFα agents. With accumulating experience, the treatment guideline for anti-TNFα therapy in latent tuberculosis is now well established. It is noteworthy that there are a number of case reports describing hepatitis B virus (HBV) reactivation in otherwise asymptomatic carriers who received anti-TNFα treatment. Anti-TNFα agents are now utilized as a promising treatment regimen for RA and AS treatment for even HBsAg carriers, yet there are still concerns of the risk of anti-TNFα therapy contributing to HBV reactivation. In our previous studies, we found that anti-viral therapy before starting anti-TNFα treatment may reduce the incidence of HBV reactivation, and that entecavir is likely more suitable in long-term prophylaxis for HBsAg carriers under anti-TNFα treatment. This justifies the need of a prospective trial that could demonstrate the long-term effects of prophylaxis in using anti-TNFα therapy in this subgroup of patients. It would help clinicians understand 1) whether anti-viral therapy is necessary in inactive HBsAg carriers initiating anti-TNFα treatment, and 2) at what time point would we most likely witness HBV reactivation after starting anti-TNFα therapy without anti-viral therapy coverage. In addition to established nationwide network of Rheumatologists working in major academic institutes in Korea, our division in Seoul National University Hospital has led many multi-center trials throughout the past years. In summary, the question of whether to combine anti-viral prophylaxis in HBsAg carriers starting anti-TNFα therapy is an important issue to Rheumatologists. There is no guideline for managing this subset of patients, and clinicians normally begin anti-viral therapy after the patient's liver function worsens. Therefore, our nationwide network of specialists proposes to launch a prospective study to investigate the benefit of anti-viral prophylaxis with entecavir in HBsAg carriers starting anti-TNFα treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis B, inactive HBsAg carriers or anti-HBc antibody positive patients with AST, ALT level equal or lower than 2x ULN
* Patient who has systemic rheumatic disease for which anti-TNFα treatment indication has been approved by the KFDA; rheumatoid arthritis (RA, 1987 ACR criteria), ankylosing spondylitis (AS, modified New York criteria), psoriatic arthritis (PsA, modified ESSG criteria), and juvenile rheumatoid arthritis (JRA, 1977 ACR criteria).
* Patient who is eligible to start anti-TNFα treatment (etanercept, infliximab, adalimumab, golimumab, and certolizumab pegol) due to treatment failure of other DMARDs against underlying RA, AS, PsA, or JRA. Patient who also fully understands that anti-TNFα agent expenses are not covered in this study.
* Patient who is willing and able to comply with the study drug regimen and all other study requirements
* Patient who is willing and able to provide a written informed consent to participate in the study

Exclusion Criteria:

* Patient who has liver cirrhosis or a history of hepatocellular carcinoma (HCC) or findings suggestive of HCC, such as suspicious foci or elevated serum alpha fetoprotein (AFP)
* Patient who received interferon or other immunomodulatory treatment for HBV infection in the 12 months before screening for this study
* Patient who has concomitant other chronic viral infection (HCV or HIV)
* Patient who is pregnant or breastfeeding or willing to be pregnant
* A history of chronic infection, recent serious or life-threatening infection. Especially,

  * Patient with current clinical or laboratory evidence of active tuberculosis (TB) or latent TB unless there is documentation of prior anti-TB treatment was appropriate in duration according to the Korea Food and Drug Administration (KFDA) guidelines for management of latent TB in patients being treated with biologic agents
  * Patient with a history of herpes zoster within 2 months before screening for this study
* Active malignancy or a history of treated malignancy less than 5 years prior to screening
* Patients who are not cooperative or unable to comply with the study procedures
* Patients with any other condition which the investigator's judgment would make the patient unsuitable for inclusion in the study such as alcohol and drug abuse

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
The frequency (events) of HBV reactivation | 48 weeks
  1. Elevated HBV DNA titer: ≥1 log10 rise in HBV DNA level compared with baseline level (virologic breakthrough), along with
  2. Increase of AST or ALT above 32 x upper limit of normal (ULN) (biochemical breakthrough)

SECONDARY OUTCOMES:
Incidence of HBV reactivation among different anti-TNFα treatment groups | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yeong wook Song, MD, PhD, Principal Investigator — Division of Rheumatology, Seoul National University Hospital
Locations (22):
- South Korea (22):
  - Hallym University Sacred Heart Hospital, Anyang
  - Dong-A University, College of Medicine, Busan
  - Daegu Catholic Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejun
  - Daejun Eulji University Hospital, Daejun
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Seoul National University Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Konkuk University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Gangdong Hospital, Seoul
  - Kyunghee University Medical Center, Seoul
  - Severance Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - Ajou University Hospital, Suwon